CLINICAL TRIAL: NCT07213713
Title: Evaluation of Anti-Xa Activity in Patients With Severe Obesity After Subcutaneous Injection of Enoxaparin for Antithrombotic Prophylaxis at Two Different Sites.
Acronym: EPOS
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Candia Erica, Prof.ssa Erica De Candia, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7741
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Venous Thromboembolism; Obese Patients
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate appropriateness of enoxaparin bioavailability at two different sites of subcutaneous administration (arms or abdomen) in primary or secondary prevention of thromboembolism in a population of patients with severe obesity

ELIGIBILITY:
Inclusion Criteria:• age >18 years,

* BMI >40 kg/m2
* indication to primary or secondary thromboprophylaxis (Padua Score > 4), as clinical practice

Exclusion Criteria:• indication to full dose anticoagulant,

* creatinine clearance <30 mL/min (based on Cockcroft-Gault equation using adjusted body weight),
* pregnant women,
* low platelet count (<50.000/microL or <100.000/microL plus additional risk factors for bleeding),
* active bleeding,
* active gastroduodenal ulcer,
* severe bleeding diathesis,
* recent/planned/emergency high bleeding-risk surgery/procedure,
* major trauma,
* acute intracranial hemorrhage,
* bleeding within the three months prior to admission,
* known hypersensitivity to enoxaparin (e.g. pruritus, urticaria, anaphylactic/anaphylactoid reactions),
* history of immune mediated heparin-induced thrombocytopenia (HIT),
* severe uncontrolled hypertension,
* diabetic or hemorrhagic retinopathy,
* concurrent administration of subcutaneous drugs (i.e. insulin, GLP-1 receptor agonists, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational study, multicentric. Target population: Patients with BMI 40 kg/m2 hospitalized, candidates for anticoagulation therapy in prophylaxis (PADUA score 4).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the achievement of both target anti-factor Xa levels at peak, defined as 0.2 to 0.4 IU/mL, and at trough, defined as >0.1 IU/mL. | 24 months
  To evaluate appropriateness of enoxaparin bioavailability at two different sites of subcutaneous administration (arms or abdomen) in primary or secondary prevention of thromboembolism in a population of patients with severe obesity

IPD SHARING:
Plan to Share IPD: No